CLINICAL TRIAL: NCT02041247
Title: Assessment of VAC-3S Therapeutic Properties When Combined With Standard Antiretroviral Therapy (ART) in the Course of HIV-1 Infection. A European, Randomized, Double Blind Placebo-controlled Phase II Study
Brief Title: Assessment of VAC-3S Therapeutic Properties When Combined With Standard ART in the Course of HIV-1 Infection
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: InnaVirVax (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IPROTECT1; 2013-002735-23 (EudraCT Number)
Record Dates: First submitted 2013-11-27; First posted 2014-01-22 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-06

CONDITIONS: HIV

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- VAC-3S 16µg/administration (Active Comparator): VAC-3S 16µg/ml administered every 4 weeks for 3 months followed by 3 maintenance vaccinations every 12 weeks after the third initial vaccination.
  Interventions: Biological: VAC-3S
- VAC-3S Placebo (Placebo Comparator): VAC-3S placebo administered every 4 weeks for 3 months followed by 3 maintenance vaccinations every 12 weeks after the third initial vaccination.
  Interventions: Biological: VAC-3S
- VAC-3S 32 µg/administration (Active Comparator): VAC-3S 32µg/ml administered every 4 weeks for 3 months followed by 3 maintenance vaccinations every 12 weeks after the third initial vaccination.
  Interventions: Biological: VAC-3S
- VAC-3S 64 µg/administration (Active Comparator): VAC-3S 64µg/ml administered every 4 weeks for 3 months without maintenance vaccination.
  Interventions: Biological: VAC-3S

INTERVENTIONS:
Biological: VAC-3S — VAC-3S is administered via intra-muscular route in the arm.

SUMMARY:
The purpose of this study is to evaluate the protective effect of VAC-3S in controlled HIV patients receiving standard of care antiretroviral treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Documented HIV-1 infection,
2. Adults > 18 and < 60 years of age,
3. Able and willing to comply with the protocol, including availability for all scheduled study visits,
4. Provided a signed written informed consent,
5. Meets study screening physical, medical history and laboratory assessments (defined below),
6. On stable antiretroviral therapy that is consistent with the current standard of care for at least 12 months prior to study screening,
7. Plasma HIV RNA < 50 cps/mL during the previous 12 months,
8. CD4+ T cell count at screening > 200 and < 500 cells/mm3,
9. Adequate hematology, biochemistry, and metabolic blood tests defined as being less than grade 2 according to the Division of AIDS Adverse Events (See Appendix 23.1), except for the numeration of CD4 and for the numeration of lymphocytes,
10. Adequate hepatic and renal function defined as being less than Grade 2 according to the Division of AIDS Adverse Events (See Appendix 23.1),
11. Female patients of childbearing age with one documented negative blood pregnancy tests between Screening and Visit 1/Month 0; Female patient of childbearing potential must be receiving two forms of effective contraception and must be willing to use them throughout the study duration. These include oral, transdermal, systemic or implant contraception birth control, intra-uterine devices (IUD), abstinence and double barrier method such as diaphragm with spermicidal gel or other recommended double barrier method,
12. Affiliated with the National Medical Insurance System,
13. Believed by investigator to be able and willing to comply with the requirements of the study protocol and will be available for all scheduled visits at the study site.

Exclusion Criteria:

1. Not meeting all of the inclusion criteria listed above,
2. Administration of any investigational drug or device within 28 days prior to screening,
3. Prior history of an AIDS-defining event in the past 5 years,
4. Active co-infection with either Hepatitis C Virus (HCV) or Hepatitis B Virus (HBV) or any other active viral hepatitis co-infection,
5. Any acute or clinically significant infections within the past month,
6. Known allergy or intolerance to components of VAC-3S as documented through medical records or via patient interview,
7. Chronic active liver disease as documented by any of the following laboratory assessments: ultrasound, clinical assessment, liver biopsy or equivalent non-invasive methods,
8. Receipt of any known vaccinations within the past 1 month prior to screening,
9. Receipt of any agent in the past 12 months that exerts a known immunological effect (e.g. includes but not limited to IL-2, IL-7, growth hormone…),
10. Patients with Insulin Dependent Diabetes Mellitus, patients receiving anti-diabetic treatment, anticoagulants (excluding daily "baby-dose" aspirin) or daily NSAIDs within one week of study enrollment,
11. Receipt of any contraindicated medications listed in Appendix 23.2,
12. History of or active auto-immune disease,
13. Acute or chronic psychiatric conditions which in the opinion of the investigator would need continual psychological support and/or medications incompatible with study participation,
14. Patients with contraindications to intramuscular injections including, but not limited to, patients with thrombocytopenia and/or anomalies of the coagulation system,
15. Any uncontrolled chronic or acute condition that in the opinion of the investigator would compromise safety of the patient or the ability to properly administer the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-09 (Actual); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
anti-3S antibodies titer | From D0 to week 24

SECONDARY OUTCOMES:
tolerance to 6 vaccinations of VAC-3S | From D0 to week 72
  safety parameter changes according to the DAIDS (Division of Acquired Immunodeficiency Syndrome) adverse events (AEs) grading table.Safety parameters include adverse events, vital signs, physical examinations, laboratory tests (hematology, blood chemistry, viral load, CD4 and CD8 counts)
blood inflammatory marker concentrations | From D0 to week 72
  Inflammatory markers include: Highly sensitive C-reactive protein (hsCRP), Highly sensitive Recombinant human interleukin 6 (hsIL-6), Soluble CD14 (sCD14), Soluble CD163 (sCD163), D-dimer, Interferon (IFN)-gamma inducible protein 10 (IP-10), Tumor necrosis factor receptor 1 (sTNFR1) and 2 (sTNFR2), Immunoglobulin G (IgG),
immunogenic characteristics of VAC-3S | From D0 to week 72
  anti-3S antibody titers and determination of anti-3S antibody isotypes and avidity
lymphocyte phenotype markers | From D0 to week 72
  Phenotype markers include: Nkp44L expression on the surface of CD4+ T lymphocytes, phenotypic markers of of lymphocyte differentiation and activation
secondary virological effects | From D0 to week 72
  3S gp41 sequences and proviral HIV reservoir

CONTACTS AND LOCATIONS:
Overall Officials: Raphael Ho Tsong Fang, DVM PhD, Study Director — InnaVirVax
Locations (12):
- France (9):
  - Hôpital Sud Francilien, Corbeil-Essonne
  - Hôpital de la Croix Rousse, Lyon
  - Hôpital Gui de Chauliac, Montpellier
  - Hôpital Saint-Antoine, Paris
  - Hôpital Pitié Salpêtrière, Paris
  - Hôpital Cochin Saint Vincent de Paul, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Hôpital Bichat - Claude Bernard, Paris
  - Hôpital Tenon, Paris
- Germany (2):
  - Jürgen Rockstroh, Bonn
  - Gerd Fätkenheuer, Cologne
- Hospital Clinic University of Barcelona, Barcelona, Spain